CLINICAL TRIAL: NCT02093455
Title: Effects of Chardonnay Seed Flour on Vascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Whole Vine Products (Unknown)
Responsible Party: Principal Investigator, Amir Lerman, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-007023
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: 1. Endothelial Dysfunction (EndoPAT Score <=2)
Keywords: Endothelial function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chardonnay Seed Flour (CSF) (Active Comparator): Prepackaged capsules taken 3 times per day. During the first month, the total dose will be 15 g/d. For months 2-4, the total dose will be 30 g/d.
  Interventions: Dietary Supplement: Chardonnay Seed Flour (CSF)
- Placebo (Placebo Comparator): Pre-packaged capsules taken 3 times per day. For the first month, a total of 15 g/d. During months 2 - 4, a total of 30 g/d.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Chardonnay Seed Flour (CSF) — CSF is made from wine grape skins and seeds.
  Arms: Chardonnay Seed Flour (CSF)
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded trial (Chardonnay seed flour vs. placebo - in pill form) with the purpose to test the impact of a four-month supplementation with Chardonnay Seed Flour (CSF) on endothelial function. Chardonnay flour is made from wine grape skins and seeds. We will examine the effect of CSF on parameters such as endothelial function (via EndoPAT testing), plasma lipid levels, glucose tolerance, insulin resistance, inflammatory markers, oxidative stress surrogates, endothelial progenitor cells (EPCs) as well as the makeup of and impact on the gut microbiome (via stool samples).

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years old
2. Demonstrated endothelial dysfunction (EndoPAT score <= 2) at time of screening.

Exclusion criteria:

1. Age below 18 or above 80
2. Endothelial function greater than 2.0 at baseline
3. Hypertension (at screening): any patient with systolic blood pressure (SBP >=170 mmHg or diastolic blood pressure >= 110 mmHg, or hypotension (SBP < 100 mmHg
4. Abnormal liver function tests
5. Uncontrolled Diabetes Mellitus or the use of metformin for Diabetes Mellitus
6. Difficulty swallowing capsules
7. Gastrointestinal disease manifesting with symptoms of malabsorption such as celiac disease or Crohn's disease
8. Non-English speakers
9. Vulnerable populations unable to consent such as prisoners or dependents
10. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the CSF including, but not limited to, any of the following:

    1. History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy or bowel resection
    2. Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase
    3. Evidence of hepatic disease as determined by a history of hepatic encephalopathy, a history of cirrhosis, esophageal varices, or a history of portocaval shunt.
11. History of hypersensitivity to any of the study supplement or suspected contraindications to the study supplement.
12. History of noncompliance to medical regimens or unwillingness to comply with the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-03; Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Endothelial function as measured by reactive hyperemia EndoPAT scores | Baseline to 4 months
  Endothelial function (Endothelial Peripheral Arterial Tonometry - EndoPAT) Testing will generate a score at baseline that will be compared to a second EndoPAT test which will be conducted again after the study subjects have taken the study product for 4 months. These scores will be used to determine if the study product had an effect on endothelial function.

SECONDARY OUTCOMES:
Change in High Sensitive C-reactive protein (hsCRP) | Baseline to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Corban MT, Widmer RJ, Cilluffo R, Kazeck MA, Lennon RJ, Lerman LO, Lerman A. The effect of polyphenol-rich chardonnay seed supplements on peripheral endothelial function. Eur J Nutr. 2020 Dec;59(8):3723-3734. doi: 10.1007/s00394-020-02203-6. Epub 2020 Feb 17. PMID 32067098
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials